CLINICAL TRIAL: NCT04916704
Title: Subclinical Cytomegalovirus Reactivation in Patients With Newly Diagnosed or Relapsed ANCA-associated Vasculitis and Adverse Clinical Outcomes
Brief Title: Subclinical Cytomegalovirus Reactivation in Acute ANCA-associated Vasculitis
Acronym: REACTIVAS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dimitrios Chanouzas, Consultant Nephrologist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: 294850
Record Dates: First submitted 2021-05-18; First posted 2021-06-07 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: ANCA Associated Vasculitis
Keywords: CMV reactivation; ANCA associated vasculitis; CD4+CD28null T-cells; Infection; Immunosuppression
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will collect blood and urine samples. Blood will be processed to derive peripheral blood mononuclear cells (PBMC), PBMC pellets to allow DNA isolation and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMV seropositive: New diagnosis of AAV as evidenced by relevant biopsy and / or clinical diagnosis in the context of a positive ANCA antibody OR major relapse of previously diagnosed AAV that requires re-induction of remission treatment with intravenous rituximab or cyclophosphamide together with high dose oral corticosteroids. CMV IgG positive.
- CMV seronegative: New diagnosis of AAV as evidenced by relevant biopsy and / or clinical diagnosis in the context of a positive ANCA antibody OR major relapse of previously diagnosed AAV that requires re-induction of remission treatment with intravenous rituximab or cyclophosphamide together with high dose oral corticosteroids. CMV IgG positive. CMV IgG negative.

SUMMARY:
This is a prospective observational study to determine the frequency and magnitude of Cytomegalovirus (CMV) reactivation in patients with anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitides (AAV) in the acute phase of the disease (within 12 months of diagnosis or relapse and commencement of induction of remission therapy) and its association with clinical outcomes. The investigators will also explore whether CMV reactivation causes an increase in CCR2 expressing monocytes, and whether these monocytes cause persistent kidney damage in AAV.

The investigators hypothesise that reactivation of CMV during the initial 12 months following diagnosis or relapse of AAV occurs frequently but is generally asymptomatic. Based on the investigators' preliminary data the investigators further hypothesise that subclinical reactivation of CMV during this period will be associated with adverse clinical outcomes, including the severity of vasculitis, the response to treatment and the damage caused by vasculitis. Finally, they hypothesise that subclinical CMV reactivation leads to amplification of renal damage in AAV through a monocyte CCR2/CCL2 driven pathway.

The investigators' research has recently shown that asymptomatic reactivation of CMV is a frequent event in AAV patients, occurring in roughly 25% of AAV patients in remission. However, the frequency of asymptomatic reactivation of CMV during the acute phase of the disease is not known. The investigators have previously shown that CMV infection and surrogate markers of CMV reactivation in patients with AAV are associated with worse outcomes such as reduced kidney function, increased risk of infection and death, increased risk of blood clots and increased stiffness of the blood vessels, which is a risk factor for heart disease and stroke. The investigators also have preliminary findings suggesting that in patients with AAV and CMV reactivation, the more CCR2 expressing monocytes in the blood, the worse the kidney function. If CMV reactivation during the acute phase of the disease is common and linked with worse outcomes, this study may then lead on to future research involving treatment to prevent CMV reactivation aiming to improve patient outcomes.

The investigators will be looking to recruit patients under the care of the Queen Elizabeth Hospital with newly diagnosed or recently relapsed AAV in the last 2 weeks who are positive for previous CMV infection.The investigators will follow these patients up with 10 visits over 12 months; where possible these will coincide with participants' usual vasculitis clinic appointments. At each visit the participants will be required to give blood and urine samples and answer questions related to their vasculitis. Kidney biopsy tissue taken at diagnosis will be used to assess mechanisms of injury during CMV reactivation.

DETAILED DESCRIPTION:
INTRODUCTION/BACKGROUND:

This is an observational study to determine the frequency and magnitude of CMV reactivation in patients with AAV in the acute phase of the disease (within 12 months of diagnosis or relapse and commencement of induction of remission therapy).

AAVs are systemic autoimmune inflammatory conditions characterized by necrotising inflammation affecting small to medium blood vessels leading to end-organ damage. Without treatment AAV is life-threatening; treatment involves powerful immunosuppression to induce remission, followed by maintenance treatment to prevent disease relapse. Treatment induction for both new-onset AAV and major life-threatening relapses is usually in the form of corticosteroids in combination with either cyclophosphamide or rituximab. Whilst prognosis has significantly improved with current treatment options for AAV, there remains significant morbidity and mortality associated with these conditions, especially during the first 12 months following diagnosis and commencement of induction of remission therapy. Infection is the leading cause of death within the first 12 months, accounting for approximately 50% of mortality as well as considerable morbidity and hospitalisation.

Cytomegalovirus (CMV) is a widely prevalent herpesvirus that is not cleared after primary infection and establishes a state of persistent infection. CMV is present in over half the population by middle age and is thought to undergo a state of latency with intermittent periods of viral reactivation. This can be a significant clinical problem amongst patients that receive immunosuppression for bone marrow or solid organ transplants. Although, patients with AAV are heavily immunosuppressed, symptomatic CMV disease is uncommon in this patient group (2%). However, asymptomatic reactivation is not uncommon. In a proof-of-concept study, the investigators have shown that asymptomatic subclinical reactivation of CMV is a frequent event amongst patients with stable AAV in remission, occurring in approximately 1 in 4 CMV seropositive AAV patients in remission over a 12-month period. The investigators and others have shown that asymptomatic CMV infection is associated with key adverse clinical outcomes amongst patients with AAV, such as reduced kidney function, increased risk of infection and mortality, increased risk of venous thromboembolism, and increased arterial stiffness, a marker of cardiovascular mortality.

The investigators have previously demonstrated that subclinical reactivation of CMV is associated with the expansion of a cytotoxic T-cell subset known as CD4+CD28null T-cells. Importantly, significant expansion of CD4+CD28null T-cells is exclusively seen in CMV seropositive patients. The investigators recently demonstrated that CD4+CD28null T-cells expansion is linked to a reduced functional capacity of the CD4 compartment and subsequent reduced response to the pneumonia vaccine, amongst patients with AAV in remission. Importantly, the investigators found that participants with evidence of subclinical CMV reactivation during the 6 months preceding the vaccination did not mount a response to the vaccine, but treatment with antiviral Valacyclovir suppressed CD4+CD28null T-cells expansion and suppression of CD4+CD28null T-cells was in itself associated with a better response to pneumococcal vaccination.

The investigators anticipate that CMV reactivation will be significantly higher during the acute phase of the disease process, both with de-novo disease and major relapses, at a time where patients are exposed to intensive immunosuppressive therapy and heightened inflammation. However, the degree to which subclinical reactivation of CMV occurs during the acute phase of AAV is not currently known.

The mechanism of CMV-induced kidney damage is not yet known. The investigators have developed preliminary unpublished data that has led them to hypothesise that subclinical CMV reactivation may amplify renal injury in AAV via the expansion of CCR2 expressing pro-inflammatory monocytes. These preliminary findings suggest that in these patients, the more CCR2 expressing monocytes in the blood, the worse the kidney function. There is also an increasing amount of evidence now that blocking CCR2 monocytes in mice reduces kidney damage across a wide variety of kidney conditions. This suggests that this monocyte-induced kidney damage pathway is not just limited to patients with vasculitis and this research could be relevant to other inflammatory renal conditions.

RATIONALE:

If this current proposed study confirms that subclinical CMV reactivation occurs frequently during the acute phase of AAV and is linked to worse patient outcomes, the investigators would propose that suppression of CMV during the acute phase of the disease would be a potentially valuable therapeutic target to improve patient outcomes and will seek funding for a multi-centre interventional study to test this hypothesis.

Another important aim of this study is to investigate the contribution of monocyte induced renal damage in AAV via the CCR2 / CCL2 axis and to determine whether repeated rounds of CMV reactivation drive expansions of CCR2 monocytes that amplify renal injury. The investigators anticipate that this will be highly relevant to other conditions where there is intra-renal inflammation. The findings of this present study may facilitate patient selection for clinical trials to maximise the benefit of CCR2 blockade treatment approaches as well as open new exciting therapeutic opportunities in AAV and other renal conditions, including diabetic kidney disease.

DESIGN:

Up to 50 CMV seropositive and 20 CMV seronegative participants will be recruited within 14 days of disease presentation or major disease relapse and commencement of induction of remission therapy, over a period of 18 months. For the purposes of this study, a major relapse will be defined as a disease relapse that requires re-induction of remission therapy with high dose corticosteroids AND either rituximab or cyclophosphamide.

Study participants will be followed up for a total of 12 months during their usual clinical visits at the NIHR / Wellcome Trust Clinical Research Facility (WTCRF) at University Hospitals Birmingham NHS Foundation Trust (UHBFT). Some study visits may be conducted at a remote offsite location in order to minimize patient hospital visits in light of the current COVID-19 pandemic. It is estimated that the study will take 36 months to complete.

OBJECTIVES:

Aim 1:

To determine the frequency and clinical importance of CMV reactivation during the acute phase (first 12 months) following diagnosis or relapse of AAV and commencement of induction of remission therapy

Blood and urine samples will be drawn at all time points to measure CMV viral DNA copies by quantitative PCR.

This will be performed at UHBFT virology laboratory using a validated commercial assay, which is routinely utilized for clinical samples. As this test does not form part of standard of care for these patients, the CMV PCR results will be held back by the Virology Laboratory and released to the research team at the end of the study. The investigators will therefore be blind to the frequency of subclinical CMV reactivation over the 12-month study period whilst the clinical outcome data is collected.

In cases where there is clinical suspicion of symptomatic CMV reactivation or CMV end-organ disease, separate relevant samples will be sent as per clinical need. Should symptomatic CMV reactivation or CMV end-organ disease be diagnosed or strongly suspected, the management will be as per standard clinical practice.

Subclinical asymptomatic CMV reactivation will be defined as a detectable viral titre of > 20 copies / ml in at least one sample of blood or urine in the absence of symptoms or signs in keeping with CMV disease, and in the absence of symptoms or signs of what would be consistent with CMV syndrome (CMV syndrome as defined in the transplant population). Patients with symptomatic CMV reactivation and / or CMV end-organ disease would be excluded from these comparisons. However, based on clinical experience, the investigators anticipate that such symptomatic disease will be very uncommon in this population.

Associations between subclinical asymptomatic CMV and the following outcomes will be assessed:

* Clinical vasculitis outcomes: Birmingham Vasculitis Activity score (BVAS), time to achieve disease remission, proteinuria (urine albumin creatinine ratio), kidney function, time to renal recovery, C-reactive protein (CRP) concentration and concentration of urinary markers of inflammation (MCP-1, CD163)
* Disease damage: Vasculitis Damage Index (VDI) at 12 months
* Patient well-being: Patient-reported outcome using AAV-PRO at 12 months
* Frailty measures: frailty index, Short physical performance battery (SPPB) and hand grip strength at 12 months
* The incidence of non-CMV infections over the 12-month study period
* The immune response to clinically indicated vaccinations
* The concentration of plasma markers of inflammation, endothelial damage, and pro-coagulant activity

Disease activity will be monitored using the BVAS at all time points. Inflammation will be assessed by CRP determination at all time points (as per standard of care). Disease burden will be assessed using the VDI score at baseline, 6 and 12 months. Patient well-being will be assessed as a patient-reported outcome using the AAV-PRO tool at 0, 3 and 12 months. Clinical assessment and standard of care clinical blood and urine test monitoring will take place at all time points to evaluate disease remission, ongoing activity and document renal function, renal replacement therapy status and albumin creatinine ratio (ACR) to assess the level of proteinuria. Time to remission will be defined as time to attaining a BVAS score of 0. Time to renal recovery will be defined as time to achieving dialysis independence or time to stabilisation of renal function following initial improvement.

The concentration of urinary soluble CD163 and MCP-1 has recently been shown to accurately reflect the presence of subtle active renal vasculitis. Urinary CD163 and MCP-1 will be assessed at baseline, 3, 6, 10 and 12 months from cryopreserved urine samples.

Frailty will be assessed using the SPPB, as a global assessment of function and cognition, and hand grip strength. The SPPB will be performed at study visits at baseline, month 1 and month 12. Hand grip strength will be measured using a hand-held dynamometer at the same points. A frailty index will be calculated at the same time points, using at least 20 different deficit variables, including the SPPB, hand grip strength and questions and blood tests taken during each study visit.

Participants will be assessed at every study visit as per standard of care and any infection experienced by the participants will be documented along with treatment received. Participants will be vaccinated with clinically indicated vaccinations as per standard of care during the follow up period. A plasma sample will be drawn immediately prior to vaccination and 2 months after vaccination to measure vaccination specific functional antibodies in order to determine the response to vaccination. Samples will be tested at the Clinical Immunology Laboratory (University of Birmingham), using a validated assay utilized for clinical samples.

Plasma and peripheral blood mononuclear cells (PBMC) will be collected from participants at the specified time points outlined in Table 1 and cryopreserved.

Whole blood will be collected in EDTA tubes (4mL) and centrifuged to yield plasma. Citrated whole blood (3.5mL) will also be collected and centrifuged within 1 hour of collection to yield platelet-free plasma, before being frozen at -80 degrees Celsius until further use. Whole blood will be collected in lithium heparin tubes (42mL) and processed within four hours to separate PBMC. Whole blood will also be stained with monoclonal antibodies to enumerate peripheral blood immune subsets.

Plasma aliquots will subsequently be thawed and batch assayed to measure markers of endothelial damage and markers of inflammation and microparticle tissue factor activity. PBMC will be thawed and immunophenotyped to determine the extended immunophenotype and activation status of CD4+CD28null T-cells.

CMV seronegative patients will be used as controls for comparison of these outcome measures at 3 monthly intervals (baseline, months 3, 6, 10, 12). The same procedures will be undertaken for CMV seronegative patients, apart from assessment of CMV PCR.

Aim 2:

Characterisation of the local and systemic monocytic repertoire in relation to CMV reactivation

Flow cytometry will be used to determine the extended phenotypic profile of monocytes both in relation to CMV serostatus and viral reactivation. Furthermore, discrete monocytic subsets, initially focussing on CCR2+ and CCR2-, will be FACS-sorted and CMV viral load quantified through use of droplet digital PCR. Single cell RNA-Seq will be applied to appropriate subpopulations identified by CMV carriage. The profile and number of virally infected and CCR2+ monocytes will then be compared to episodes of CMV reactivation, to determine whether repeated rounds of CMV reactivation drives expansion of this cell subset.

Aim 3:

Assessment of potential mechanisms of renal damage induced by CCR2+ monocytes

Kidney tissue from our recruited patients, obtained at the time of diagnosis of new or relapsing disease with renal involvement from a standard of care renal biopsy, will be used to explore the relationship between CMV reactivation, monocytes and kidney damage. We anticipate the vast majority of patients with renal involvement will have a renal biopsy (50-70% of total recruited patients). Additional biopsy tissue will not be required; the cores obtained as per standard of care will be sufficient for research purposes.

Renal tissue will be analysed to determine expression of markers of interest to explore the mechanisms underlying tissue damage in renal biopsies using scanned biopsy image software. The focus will be on (i) potential anatomical sites of viral replication, (ii) phenotype and infiltration of CD4+CD28- T cells and (iii) detailed transcriptional analysis of CCR2+ monocytes. These observations will also be correlated with matched urinary MCP-1 and CSF2 concentration to determine the potential value of these as markers of intrarenal monocyte infiltration.

To further interrogate the potential mechanisms of monocyte-induced glomerular injury, in-vitro add-back experiments will determine whether CCR2 monocytes are capable of damaging glomerular endothelium.

SCHEDULE OF ASSESSMENTS:

All study participants will have a maximum of 11 interactions with the research team. The timing of the study visits has been selected to coincide with clinical visits that patients would be expected to attend as part of their ongoing clinical management.

Participants will either be recruited as in-patients or out-patients. For in-patients, the first contact will be face-to-face during their inpatient stay, to provide verbal and written information, including a Patient Information Sheet (PIS). The baseline visit will then occur at least 24 hours later, at which the patient will be given the option to be recruited to the study.

For out-patients, the first contact will be written information in the post (PIS) and contact details for the research team will be provided. This will be followed by a telephone consultation to answer any questions and establish interest. For those patients who express interest, the third point of contact (baseline visit) will be face-to-face with the research team at their routine AAV clinic appointment or treatment schedule; this will not be an additional hospital visit.

A total of 10 study clinic appointments will be held at UHBFT for CMV seropositive and 5 for CMV seronegative subjects. During the baseline visit participants will be recruited to the study either during their hospital admission or during a scheduled hospital visit either to the clinic or for treatment. After inclusion/exclusion criteria are met, written informed consent will be obtained for all patients prior to enrolment. A clinical assessment with be made, BVAS and VDI calculated, AAV-PRO completed, SPPB and hand grip strength carried out and blood and urine samples collected.

The remaining follow-up visits will be scheduled at intervals over the next 12 months. In light of the current COVID-19 pandemic, patients are only attending face-to-face hospital appointments when necessary, with telephone consultations being conducted when appropriate; decisions on who is allocated to which appointment type are being made on an individual patient basis. The investigators will not bring participants to the hospital for additional study visits where they cannot come through a 'clean' pathway; in these circumstances, with the agreement of the subject, the investigators will arrange for home study visits.

At each follow-up visit the research team will complete a clinical assessment, calculate BVAS and VDI where applicable, conduct SPPB and measure hand grip strength where applicable and further blood and urine samples will be taken. The AAV-PRO may be sent out to patients a few days prior to their study visit via the post or email (at their preference) and patients will be asked to return completed forms at their visit. The investigators will aim to give participants clinically indicated vaccinations during follow up as per standard of care at month 10; the investigators will contact the patient's GP to clarify previous vaccine history prior to administration. Participants will have completed the study when the 12-month follow-up visit has been completed.

Renal biopsy tissue obtained at the time of diagnosis of new or relapsing disease, with renal involvement, from a standard of care renal biopsy, will be used to explore the relationship between CMV reactivation, monocytes and kidney damage. We anticipate the vast majority of patients with renal involvement will have a renal biopsy (50-70% of total recruited patients). Additional biopsy tissue will not be required; the cores obtained as per standard of care will be sufficient for research purposes.

SAMPLE SIZE:

This is an observational study with the primary outcome to estimate the rate of subclinical CMV reactivation, so there is no formal power calculation. There is also a limit to the number of patients that will meet the inclusion criteria during the study timeframe. As such, no formal power calculation was performed, with the aim instead being to recruit as many patients as is feasible.

The investigators estimate that they will recruit up to 50 CMV seropositive and 20 CMV seronegative patients over 18 months, as they expect this number will be the maximum feasible within a single centre with a population of 250 patients (around 40 new diagnoses AAV/year). The investigators expect around 70% of this cohort will be CMV seropositive. Patients recruited following a major relapse of AAV will be limited to 30% of the total study population. Historically, the AAV cohort of patients is a very well-motivated group of patients with very high participation in research studies and usually excellent clinic attendance. As such, the investigators would expect the vast majority of eligible patients to be willing to join the study, and for negligible loss to follow up or study withdrawal.

STATISTICAL ANALYSIS:

Analysis of study data will be conducted by the research team with the assistance of a statistical advisor. The main analysis will be conducted on the entire study cohort, although planned sub-group analysis will also evaluate potential differences between patients with newly diagnosed AAV, and those with a major relapse of previously diagnosed disease.

Analysis of the primary outcome of CMV reactivation will be performed using a time-to-event approach, in order to account for the time that this was identified, and the potential for varying follow up times across the cohort in patients that do not complete the study. As such, patients will be censored where they are either lost to follow up, withdraw from the study, or die during the study period. In addition to performing this analysis for the cohort as a whole, a subgroup analysis will also be performed after excluding those with CMV reactivation at the baseline visit, in order to estimate the rate of new-onset CMV reactivation after the commencement of treatment for AAV.

The remaining clinical outcomes are based on comparisons between patients with asymptomatic CMV reactivation, and those without CMV reactivation, as well as between those who are CMV seropositive and those who are seronegative as a control group. Analyses will be performed which consider the actual viral titre in those where it is detectable, to assess whether there is a dose-response relationship between viral load and patient outcomes.

Analyses of the secondary and tertiary outcomes will utilise differing methodologies, depending on how the outcomes of interest are quantified. For outcomes measured at a single time point (e.g. VDI at 12 months), comparisons by CMV reactivation status will be performed using independent group comparisons, such as independent samples t-tests. Outcomes measured at multiple time points (e.g. clinical bloods recorded at every visit) will be assessed using repeated-measures analyses, in order to account for the correlations between multiple samples contributed by the same patient. For time-to-event outcomes (e.g. time to achieve disease remission), analyses will be based on Kaplan-Meier curves and Cox regression models. Finally, count-based outcomes (e.g. development of non-CMV infections) will be analysed as an incidence (per patient-year), in order to account for the follow up time contributed by each patient.

In all analyses, the asymptomatic CMV reactivation status will initially be considered as a fixed-effects variable, such that patients will be assigned to a CMV reactivation group, regardless of when this was first diagnosed. However, analyses will also be performed where this factor is treated as a time-dependent covariate, such that all patients are assigned to the negative group at the commencement of follow up, before transitioning to the CMV reactivation group at the time that this was diagnosed.

Laboratory-based outcomes focused around phenotyping and enumerating monocytes, urinary markers of interest and targets within renal tissue will involve comparisons between CMV seropositive and seronegative groups along with CMV reactivation status. Comparisons between two groups will be done by unpaired t-tests.

QUALITY ASSURANCE/MONITORING:

The study may be subject to inspection and audit by UHBFT under their remit as sponsor and other regulatory bodies, to ensure adherence to GCP and regulations. The named investigators will allow study-related monitoring, audits, Research Ethics Committee review and regulatory inspectors (where appropriate) by providing direct access to study source data and associated documents e.g. consent forms, UHBFT laboratory results etc.

ADVERSE EVENTS:

A SAE form should be completed and submitted to the Principal Investigator for all SAEs within 24 hours. The Principal Investigator's assessment of causality of SAEs (i.e. their relationship to trial treatment) will be reported on the Serious Adverse Event form; the investigators do not anticipate any related adverse events associated with this observational study. Related and/or unexpected events will be reported to the main Research Ethics Committee by the Chief Investigator within 15 days of them becoming aware of the event, in line with HRA recommendations.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of AAV as evidenced by relevant biopsy and / or clinical diagnosis in the context of a positive ANCA antibody OR major relapse of previously diagnosed AAV that requires re-induction of remission treatment with intravenous rituximab or cyclophosphamide together with high dose oral corticosteroids
* Age >18 years
* Willingness to participate in the study and attend clinic and study visits
* Able to provide written informed consent

Exclusion Criteria:

* Strong suspicion of alternative diagnosis other than AAV
* Subjects who do not have capacity to consent to study participation as defined by the Mental Capacity Act 2005
* Inability or unwillingness to attend study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with new or relapsing AAV will be identified through the vasculitis multi-disciplinary weekly meeting, clinician colleagues and the vasculitis specialist nurse. Up to 70 participants (50 CMV seropositive and 50 CMV seronegative) will be recruited within 14 days of disease presentation or major disease relapse and commencement of induction of remission therapy, over a period of 18 months. For the purposes of this study, a major relapse will be defined as a disease relapse that requires re-induction of remission therapy with high dose corticosteroids AND either rituximab or cyclophosphamide.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of CMV reactivation during the acute phase (first 12 months) following diagnosis or relapse of AAV and commencement of induction of remission therapy | This will be assessed at month 12 (end of study)
  As assessed by measurable viral load (titre >20 viral copies/ml) on quantitative PCR assessment of any blood or urine sample during the 12 month study period

SECONDARY OUTCOMES:
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and Birmingham Vasculitis Activity Score (BVAS) | This will be assessed at day 0, day 14, month 1, 2, 3, 4, 5, 6, 10 and 12.
  The correlation between subclinical CMV reactivation during the acute phase of AAV and BVAS across the study period
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and time to achieve disease remission | This will be assessed at day 0, day 14, month 1, 2, 3, 4, 5, 6, 10 and 12 to identify disease remission
  Time to achieve disease remission (defined as a BVAS score of 0)
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and urine albumin creatinine ratio (ACR) at 12 months | This will be assessed at month 12.
  The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and urine albumin creatinine ratio (ACR) at 12 months
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and renal function at 12 months | This will be assessed at month 12.
  Serum creatinine will be used to measure renal function
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the time to renal recovery | This will be assessed at day 0, day 14, month 1, 2, 3, 4, 5, 6, 10 and 12 to identify renal recovery
  The time to renal recovery will be defined as time to achieving dialysis independence or time to stabilisation of renal function (measured in days)
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the Vasculitis Damage Index (VDI) at 12 months | This will be assessed at month 12
  The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the Vasculitis Damage Index (VDI) at 12 months
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and patient well-being | This will be assessed at month 3 and month 12
  This is a patient-reported outcome using AAV-PRO tool
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the concentration of plasma CRP across the study period | This will be assessed at day 0, day 14, month 1, 2, 3, 4, 5, 6, 10 and 12
  The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the concentration of plasma CRP across the study period
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the concentration of urinary MCP-1 and CD163 across the study period | This will be assessed at day 0, day 14, month 1, 2, 3, 4, 5, 6, 10 and 12
  The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the concentration of urinary MCP-1 and CD163 across the study period
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and frailty | This will be assessed at day 0, month 1 and month 12
  A frailty index will be calculated at the same time points, using at least 20 different deficit variables, including the SPPB (scored 0-12), hand grip strength (highest measurement of 3 on each hand) and questions and blood tests taken during each study visit. These outcome measures will be combined to create an overall frailty score.
The correlation between subclinical asymptomatic CMV reactivation during the acute phase of AAV and the incidence of non-CMV infections over the 12-month study period | This will be assessed at day 0, day 14, month 1, 2, 3, 4, 5, 6, 10 and 12
  Participants will be assessed at every study visit and any infection experienced by the participants will be documented in a questionnaire along with treatment received. This will calculate an incidence of infection during the first 12 months.
The correlation between subclinical CMV reactivation during the acute phase of AAV and the antibody response ratio following clinically recommended vaccinations at 8 weeks post-vaccination | Participants will be vaccinated with clinically indicated vaccinations as per standard of care at month 10. A plasma sample will be drawn immediately prior to vaccination and 2 months after vaccination (month 12)
  The antibody response ratio is the antibody titre at 8 weeks post-vaccination / antibody titre prior to vaccination
The correlation between subclinical CMV reactivation during the acute phase of AAV and the concentration of plasma markers of inflammation | This will be assessed at baseline, month 3, 6, 10 and 12
  Plasma will be collected from participants at the specified time points during follow up to measure the concentration of TNF, IFN, IL-6 and IP-10 using ELISA.
The correlation between subclinical CMV reactivation during the acute phase of AAV and the concentration of plasma markers of endothelial damage | This will be assessed at baseline, month 3, 6, 10 and 12
  Plasma will be collected from participants at the specified time points during follow up. Elisa assays will be used to measure the concentration of Fractalkine, VCAM-1, ICAM-1, MCP-1 and P-selectin.
The correlation between subclinical CMV reactivation during the acute phase of AAV and the concentration of plasma markers of pro-coagulant activity | This will be assessed at baseline, month 3, 6, 10 and 12
  Plasma will be collected from participants at the specified time points during follow up. Elisa assays will be used to measure the concentration of Tissue Factor.

OTHER OUTCOMES:
The correlation between subclinical CMV reactivation during the acute phase of AAV and the proportion and phenotype of pro-inflammatory peripheral blood T-cell and monocyte subsets | This will be assessed at baseline, month 3, 6, 10 and 12
  Peripheral blood mononuclear cells (PBMC) will be immunophenotyped to enumerate T-cell and monocyte subsets including CD4+CD28null T-cells and CCR2 expressing monocytes at at the specified time points during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Chanouzas, MBChB, PhD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan MD, Pachnio A, Begum J, Roberts D, Rasmussen N, Neil DA, Bajema I, Savage CO, Moss PA, Harper L. CD4+CD28- T cell expansion in granulomatosis with polyangiitis (Wegener's) is driven by latent cytomegalovirus infection and is associated with an increased risk of infection and mortality. Arthritis Rheum. 2011 Jul;63(7):2127-37. doi: 10.1002/art.30366. PMID 21437878
- [Background] Chanouzas D, Sagmeister M, Dyall L, Sharp P, Powley L, Johal S, Bowen J, Nightingale P, Ferro CJ, Morgan MD, Moss P, Harper L. The host cellular immune response to cytomegalovirus targets the endothelium and is associated with increased arterial stiffness in ANCA-associated vasculitis. Arthritis Res Ther. 2018 Aug 29;20(1):194. doi: 10.1186/s13075-018-1695-8. PMID 30157919
- [Background] Chanouzas D, Sagmeister M, Faustini S, Nightingale P, Richter A, Ferro CJ, Morgan MD, Moss P, Harper L. Subclinical Reactivation of Cytomegalovirus Drives CD4+CD28null T-Cell Expansion and Impaired Immune Response to Pneumococcal Vaccination in Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. J Infect Dis. 2019 Jan 7;219(2):234-244. doi: 10.1093/infdis/jiy493. PMID 30102389